CLINICAL TRIAL: NCT01587807
Title: A Two-part, Randomised, Placebo-controlled Study to Investigatethe Safety, Tolerability, Pharmacokinetics and Pharmacodynamicsof Single Doses of Inhaled GSK1995057 in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of Inhaled GSK1995057
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 116236; 2011-005245-13 (EudraCT Number)
Record Dates: First submitted 2012-03-29; First posted 2012-04-30 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Disorders
Keywords: Infection, Quality of Life, lung injury
MeSH Terms: conditions — Respiration Disorders; Infections; Lung Injury | interventions — GSK1995057; Bronchoalveolar Lavage

STUDY DESIGN:
Who Masked: Participant

ARMS (6):
- Cohort 1 (Experimental): single inhaled dose of GSK1995057 (dose 1) or placebo
  Interventions: Drug: GSK1995057; Drug: Placebo
- Cohort 2 (Experimental): single inhaled dose of GSK1995057 (dose 2) or placebo
  Interventions: Drug: GSK1995057
- Cohort 3 (Experimental): single inhaled dose of GSK1995057 (dose 3) or placebo
  Interventions: Drug: Placebo
- Cohort 4 (Experimental): single inhaled dose of GSK1995057 (dose 4) or placebo
  Interventions: Drug: Placebo
- Cohort 5 (Experimental): single inhaled dose GSK1995057 (dose 4) with bronchoalveolar lavage (BAL)sampling procedure conducted approximately 30 minutes post GSK1995057 dose
  Interventions: Drug: GSK1995057
- Cohort 6 (Experimental): high dose of GSK1995057 or placebo followed by an inhaled LPS challenge and BAL sampling procedure.
  Interventions: Drug: GSK1995057; Procedure: bronchoalveolar lavage; Drug: LPS; Drug: Placebo

INTERVENTIONS:
Drug: GSK1995057 — inhaled dose (volume based on cohort)
  Arms: Cohort 1; Cohort 2; Cohort 5; Cohort 6
Procedure: bronchoalveolar lavage — BAL
  Arms: Cohort 6
Drug: LPS — 50 μg
  Arms: Cohort 6
Drug: Placebo — Sucrose, glycine, sodium dihydrogen phosphate and polysorbate 80 (volume to match active dose)
  Arms: Cohort 1; Cohort 3; Cohort 4; Cohort 6

SUMMARY:
GSK1995057 is a fully human, single domain antibody directed against the TNFR1 receptor. The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of inhaled GSK1995057 in healthy subjects. The study will be in two parts. Part 1 is a single-dose escalating design of 5 sequential cohorts of healthy subjects. Part 2 is a single-dose, parallel group design comprising 2 groups of healthy subjects assessing the effect of GSK1995057 on lung inflammation following inhaled LPS challenge. Actual dose administered in Part 2 will be determined from emerging safety and PK data from Part 1 and Study TFR110951.

DETAILED DESCRIPTION:
This study will be a randomised, placebo-controlled study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of single doses of inhaled GSK1995057 in healthy subjects. The study consists of 2 parts with a total of 6 cohorts. Part 1 will be conducted singleblind and Part 2 will be conducted single-blind with restrictions (i.e. subject and investigator only). The GSK Study Team and site pharmacist will remain unblinded to treatment allocation. Cohorts 1, 2, 3 and 4 (in Part 1) will receive a single inhaled dose of GSK1995057 or placebo. Cohort 5 will receive a single inhaled dose of GSK1995057 and in addition will have a bronchoalveolar lavage (BAL) sampling procedure conducted approximately 30 minutes post GSK1995057 dose. Subjects in Cohort 6 (Part 2) will be randomised to receive a high dose of GSK1995057 or placebo followed by an inhaled LPS challenge and BAL sampling procedure. Subjects will be required to visit the clinic over the course of 28 days after their dosing period for a follow up. Further visits for immunogenicity sampling may be conducted at 56 and 84 days post-first dose for subjects who show changes indicating a positive ADA response after dosing. Doses levels stipulated within the protocol are target doses based on predictions using the PK/PD model described in Section 1.2.2 of the clinical protocol. Part 1 will commence first and following acceptable safety and tolerability data will allow initiation of Part 2. All cohorts will participate in a single study session only.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests nd cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. The investigator may discuss with GSK medical monitor as required.
* Male or female between 18 and 55 years of age inclusive: A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhoea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 MlU/ml and oestradiol less than 40 pg/ml (less than 140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method. Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until the last follow-up visit.
* Normal creatinine clearance values at screening (calculated from serum creatinine by a predicting equation using Cockcroft-Gault formula), normal serum creatinine value as defined by the local reference laboratory, normal urine microscopy and no significant proteinuria on dipstick testing.
* Body weight greater than and equal to 50 kg and BMI within the range 19 - 29.9 kg/m2 (inclusive).
* No evidence of previous or active TB infection and a negative QuantiFERON TB Gold test taken within 7 days of dosing, and negative medical history with respect to active or latent mycobacterium tuberculosis complex infection.
* Normal spirometry (FEV1 greater than and equal to 85% of predicted, FEV1/FVC ratio greater than and equal to 70%) at screening. Predictions should be according to ECCS equations, and race corrections should be made for non-caucasians.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Available to complete all study assessments.
* Subjects who are able to use the inhaler device correctly.
* Able to read, comprehend and write English at a sufficient level to complete study related materials.

Exclusion Criteria:

* A history of Hepatitis B, Hepatitis C or HIV infection and/or a positive pre-study HIV, Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities. (With the exception of known Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* History of and/or a positive test for toxoplasmosis consistent with active toxoplasmosis infection at the time of enrollment.
* A positive RT-PCR test for influenza A/B.
* Current evidence or history of an influenza-like illness as defined by fever (greater than 380C) and two or more of the following symptoms within the last 7 days: cough, sore throat, runny nose, sneezing, limb/joint pain, headache, vomiting/diarrhoea in the absence of a known cause, other than influenza.
* Corrected QT interval (QTc) >450msec.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units for males or greater than 14 units for females. One unit is equivalent to 8 g of alcohol and the following can be used as a guide: a half-pint (approximately 240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject is unwilling to abstain from alcohol consumption from 24 hr prior to dosing until discharge from the clinic, and for 24 hr prior to all other out-patient clinic visits.
* Subjects with a smoking history of greater than 5 cigarettes per day in the last 3 months (Part 1); smokers are not eligible to take part in Part 2.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2012-03-28 (Actual); Primary Completion 2012-11-19 (Actual); Study Completion 2012-11-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ascending single inhaled doses of GSK1995057 | 56 Days
  Adverse event reporting, Laboratory safety data (clinical chemistry, hematology, urinalysis), Vital signs (blood pressure, heart rate, respiration rate, body temperature), ECG monitoring, Spirometry monitoring (FEV1, FVC)
Levels and specificity of anti-GSK1995057 binding antibodies. | Up to 84 Days
  Presence of anti GSK1995057 binding antibodies. Where binding antibodies aredetected, levels and specificity of the antibodies will be evaluated
Plasma pharmacokinetics of ascending single inhaled doses of GSK1995057 | 3 days
  Plasma concentrations of GSK1995057 and derived pharmacokinetic parameters in normal healthy subjects following single administration (all except Cohort 5).
Urine pharmacokinetics of single inhaled doses of GSK1995057 | 3 Days
  Urine concentrations of GSK1995057 and derived pharmacokinetic parameters in normal healthy subjects following a single administration (Part 1, except Cohort 5).
Concentration of GSK1995057 in lung epithelial lining fluid after inhalation of a single dose | 1 Day
  Bronchoalveolar lavage (BAL) concentrations of GSK1995057 and derived lung deposition parameters in normal healthy subjects following a single administration (Cohorts 5 & 6 only). Bronchoalveolar lavage (BAL) concentrations of urea (Cohorts 5 & 6 only).
Effect of single inhaled doses of GSK1995057 on biomarkers | 3 Days
  Pharmacodynamic and immune function biomarkers in serum (these may include but are not limited to sTNFR1 (free and total) and IL-6) (all except Cohort 5).
Effect of single inhaled doses of GSK1995057 on biomarkers in BAL | 1 Day
  Bronchoalveolar lavage (BAL) neutrophil counts at 6 h post LPS exposure (Cohort 5). Other pharmacodynamic and immune function biomarkers in BAL (these may include but are not limited to TNFα and IL-6) (Cohort 5).
To explore the GSK1995057 PK-PD relationship | 1 Day
  Pharmacodynamic and immune function biomarkers in serum and BALF (these may include but are not limited to sTNFR1 (free and total) and IL-6). Bronchoalveolar lavage (BAL) concentrations of GSK1995057 and derived lung deposition parameters in normal healthy subjects following a single administration (Cohort 5 and 6 only). Bronchoalveolar lavage (BAL) concentrations of urea (Cohorts 5 and 6 only). Change from baseline in IL-8 expression in ex vivo whole blood assay (WBA).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Harrow

REFERENCES:
- [Background] Proudfoot AG, O'Kane CM, Bayliffe A, Serone AP, Bareille P, Smith SP, Brown V, Wright TJ, Chen Y, Wilson R, Cordy JC, Morley PJ, Elborn S, Hind M, Chilvers ER, Griffiths MJ, Summers C, McAuley DF . A novel TNFR1-targeting domain antibody attenuates pulmonary inflammation in a human model of lung injury, via actions on the lung micro-vascular endothelium.. American Journal of Respiratory and Critical Care Medicine. 2014;189:A6589
- [Derived] Proudfoot A, Bayliffe A, O'Kane CM, Wright T, Serone A, Bareille PJ, Brown V, Hamid UI, Chen Y, Wilson R, Cordy J, Morley P, de Wildt R, Elborn S, Hind M, Chilvers ER, Griffiths M, Summers C, McAuley DF. Novel anti-tumour necrosis factor receptor-1 (TNFR1) domain antibody prevents pulmonary inflammation in experimental acute lung injury. Thorax. 2018 Aug;73(8):723-730. doi: 10.1136/thoraxjnl-2017-210305. Epub 2018 Jan 29. PMID 29382797
- See also: Results for study 116236 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116236?search=study&search_terms=116236#rs